CLINICAL TRIAL: NCT05929053
Title: The Effect of Vaccine Education Program Based on The Integrated Change Model on Vaccine Advocacy and Vaccine Literacy: A Waitlist Randomized Controlled Trial
Brief Title: Impact of Vaccine Education Program on Vaccine Advocacy and Vaccine Literacy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Artvin Coruh University (Other)
Responsible Party: Principal Investigator, Deniz Sümeyye YORULMAZ, Principal Investigator, Artvin Coruh University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ArtvinCoruhU
Record Dates: First submitted 2023-04-24; First posted 2023-07-03 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Unrecognized Condition
Keywords: Vaccines; Immunization; Literacy; Health Literacy
MeSH Terms: conditions — Literacy

STUDY DESIGN:
Intervention Model Description: Randomization and blinding are recommended in randomized controlled studies to prevent biases and show the experiment's success (15).
  Allocation: Random assignment. Block randomization will be used in the randomization process. Randomizer.org will be used to select block combinations with eight blocks. Eligible participants will be randomly assigned to the intervention or waitlist group using the permuted block randomization method on a 1:1 basis. The waiting list group will form the second set of the research, which is planned to be attempted two months later. The participant assignment list will be generated by a non-research statistician with a random distribution sequence. Assignment confidentiality will be ensured using opaque sealed envelopes containing sequence numbers. The data analyst/statistician will be blind to the participants' group assignments.
Who Masked: Participant, Outcomes Assessor
Masking Description: Single blinding(Participant blinding) will be done; participants will not be told they are in the experimental or control group. The first researcher will invite mothers to the study, which will continue until the targeted sample number(74 participants) is reached. During the participant registration, the names and contact information of the mothers will be obtained; it will be stated that they will be contacted for the training process, that the training time may be extended, and that they will be given definite training. The second researcher in the research team will explain to the first researcher that the participants are in the experimental or control group. The mothers in the control group will be assigned to the waiting list. At the end of the study, a four-session vaccination training program will be applied to the mothers in the control group in the same way and within the same scope as the experimental group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Experiment: The Vaccine Education Program based on The Integrated Change Model will be administered to the mothers in the experimental group by the researcher. The training will take place in four sessions, one week apart, and each session will last approximately 45 minutes. The training will be carried out as group training with 4-5 people. Data collection forms will be applied before and after the program.
  Interventions: Other: Vaccine Education Program Based on Integrated Change Model
- Control-waiting list (Other): Control (waiting list): The control group of the study will be the mothers who are on the waiting list. No intervention will be made to the mothers in the control group during the education process of the experimental group. After the training process of the mothers in the experimental group is completed and the post-test data are collected, all the interventions and training will be given to the mothers in the control group.
  Interventions: Other: Vaccine Education Program Based on Integrated Change Model

INTERVENTIONS:
Other: Vaccine Education Program Based on Integrated Change Model — Vaccine Education Program Based on Integrated Change Model The training will take place in four sessions, one week apart, and each session will last approximately 45 minutes. The training will be carried out as group training with 4-5 people.

SUMMARY:
This research will be carried out as a randomized controlled study with a waitlist in parallel design to evaluate the effect of the vaccine education and vaccine advocacy program prepared according to The Integrated Change Model on the level of vaccination literacy and the transformation into vaccine advocates. Research hypothesis "H0a: Vaccine education program prepared according to The Integrated Change Model does not affect vaccine literacy, H0b: The vaccine training program prepared according to the integrated change model does not affect the concepts (information sources, intention, attitude, behavior, obstacles) in the integrated change model determined for vaccine advocacy. At the end of the training, it is thought that the mothers in the experimental group will be different from the control group regarding vaccine literacy and the vaccine advocacy concepts (information sources, intention, attitude, behavior) in the model.

DETAILED DESCRIPTION:
This research will be carried out as a randomized controlled study with a waitlist in parallel design to evaluate the effect of the vaccine education and vaccine advocacy program prepared according to The Integrated Change Model on the level of vaccination literacy and the transformation into vaccine advocates. Research hypothesis "H0a: Vaccine education program prepared according to The Integrated Change Model does not affect vaccine literacy, H0b: The vaccine training program prepared according to the integrated change model does not affect the concepts (information sources, intention, attitude, behavior, obstacles) in the integrated change model determined for vaccine advocacy. At the end of the training, it is thought that the mothers in the experimental group will be different from the control group regarding vaccine literacy and the vaccine advocacy concepts (information sources, intention, attitude, behavior) in the model.

A national study on the subject was used in calculating the study's sample size. In a study conducted in Turkey, the rate of those who were hesitant about vaccination in the families of children under five years old and the rate of rejection was found to be 19.8% (1). The sample size required to eliminate this situation with vaccine advocacy was calculated as a total of 64 individuals at 0.05 alpha and 80% power level in the Gpower program. Considering the sample losses, the sample was increased by 15% (9.6 people ~ 10 people), and a total of 74 people, 37 of which were experimental and 37 control, was determined. Mothers who applied to the Family Health Centers, which are research areas, will be evaluated according to the eligibility criteria. Then researcher (DS-Y) will obtain contact information from mothers, who met the inclusion criteria, volunteered for the study, and consented, and collect pre-test. The participants will be divided into experimental and control groups using the blind technique and block randomization. The vaccination training program prepared based on The Integrated Change Model for the mothers in the experimental group will be face-to-face training. The training will be in the form of 4 sessions (with a 1-week interval) as group training for 4-5 people, and each session will last 45 minutes on average. After the training program of the mothers in the experimental group is completed, the data collection forms will be applied again to the mothers in the experimental and control groups. After the last measurement, a 4-session vaccination training program will be applied to the mothers in the control group in the same way and within the same scope as the experimental group.

The primary outcome expected from the study is the change in mothers' vaccine literacy, vaccine advocacy intention, and vaccine attitudes.

The secondary result expected from the study is the change in mothers' knowledge of vaccination and sources of vaccination information.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for the mother

1. To be residing in Artvin city center
2. To have applied to the Family Health Center No. 1 or 2 in the city center for any reason.
3. Having at least a high school graduate education level
4. Having a child in the age range that covers the national vaccination calendar (0-13 years old)
5. Turkish - speaking
6. Being literate
7. Being 18 years or older
8. Volunteering to participate in research

Exclusion Criteria:

Exclusion criteria for the mother

1. To reside outside of Artvin city center
2. To have an education level below a high school graduate
3. Having a child not between 0-13 years old
4. Not know to speak Turkish
5. Not volunteering for research

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Mothers with 0-13-year-old children
Enrollment: 74 (Actual)
Dates: Start 2023-07-03 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Vaccine literacy | 01.08.2023-31.08.2023 (within 1 month on average)
  The primary outcome expected from the study is the change in mothers' vaccine literacy, vaccine advocacy intention, and vaccine attitudes.
  Vaccine Literacy: Vaccine Literacy Scale Vaccine Literacy Scale: The scale evaluates the level of vaccine literacy. The Vaccine Literacy Scale was developed by Ahoran et al. (2017). The scale consists of 3 sub-dimensions and 13 items: Functional, Communicative, and Critical Health Literacy. The scores of the subscales are calculated separately; therefore, the scale has no total score. Responses in each subscale are divided by the number of items to obtain a score. Lower functional health literacy scores indicate higher health literacy. Higher communicative and critical health literacy scores indicate higher health literacy. The researchers previously carried out this scale's Turkish validity and reliability study (3).
  The results will be evaluated for each participant before and after the vaccine training (within 1 month on average).
Vaccine advocacy intention | 01.08.2023-31.08.2023 (within 1 month on average)
  Vaccine Advocacy Intention: Vaccine Advocacy Intent Scale
  Vaccine Advocacy Intention: Vaccine Advocacy Intent Scale Vaccine Advocacy Intent Scale: Mothers' vaccine advocacy intent will be evaluated with the Vaccine Advocacy Intent Scale. Researchers prepared the Vaccine Advocacy Intention Scale to assess mothers' intentions to engage in vaccine advocacy. The scale is scored between 0-10 points; an increase in the total score is interpreted as an increase in vaccine advocacy intention. The aim is to evaluate quantitatively mothers' intentions to be able to do vaccine advocacy.
  The results will be evaluated for each participant before and after the vaccine training (within 1 month on average).
vaccine attitudes | 01.08.2023-31.08.2023 (within 1 month on average)
  The Public Attitude Towards Vaccination Scale-Health Belief Model (PAVS-HBM): PAVS-HBM measure the public's attitude towards the vaccine according to the health belief model. The scale consists of 26 items and five sub-dimensions: sensitivity, severity, benefits, barrier, and health responsibility. Each sub-dimension is evaluated separately. Sensitivity and severity sub-dimension has four items (lowest4, highest20 points); benefit and health responsibility sub-dimension consists of five items (lowest5, highest25 points), and the barrier sub-dimension consists of eight items (lowest8, highest40 points). While the decrease in the total score in the disability sub-dimension indicates a positive attitude. An increase in the total score in other sub-dimensions means a positive attitude (4).The results will be evaluated for each participant before and after the vaccine training (within 1 month on average).

SECONDARY OUTCOMES:
Vaccine knowledge level and sources of vaccine information | 01.08.2023-31.08.2023 (within 1 month on average)
  The secondary result expected from the study is the change in mothers' knowledge of vaccination and sources of vaccination information.
  Vaccine knowledge: Vaccine Knowledge Test Vaccine Knowledge Test: Researchers conducted Vaccine Knowledge Test by reviewing the literature to evaluate mothers' knowledge about vaccines has been prepared (5-10). In the Vaccine Knowledge Test, there are 31 questions answered as true, false, and do not know. Expert opinion was taken while creating the Vaccine Knowledge Test, and the content validity was evaluated. The lowest score that can be obtained from the Vaccine Knowledge Test is 0, and the highest score is 31; The increase in the total score indicates that the vaccination knowledge is high.
  The results will be evaluated for each participant before and after the vaccine training (within 1 month on average).
Sources of vaccine information | 01.08.2023-31.08.2023 (within 1 month on average)
  Vaccine Information Resources: Vaccine Knowledge Resources Questionnaire
  Vaccine Knowledge Resources Questionnaire: Vaccine information resources of mothers will be evaluated with the Vaccine Information Resources Questionnaire. The researchers reviewed the Vaccine Information Resources Questionnaires to determine which sources mothers used as vaccine information sources in the literature (1, 11-14). There are eight questions in this form; The questions are answered with yes or no. After the training, mothers are expected to obtain information from reliable information sources such as WHO and UNICEF.
  The results will be evaluated for each participant before and after the vaccine training (within 1 month on average).

CONTACTS AND LOCATIONS:
Locations (1):
- Deniz S. Sümeyye YORULMAZ, Merkez, Artvin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The personal information of the participants will only be used by the researchers.

REFERENCES:
- [Derived] Yorulmaz-Demir DS, Kocoglu-Tanyer D. The Effect of the Vaccine Education Program Prepared Using The Integrated Change Model on Mothers' Vaccine Advocacy and Vaccine Literacy: A Waitinglist Randomized Controlled Trial. J Pediatr Health Care. 2025 May-Jun;39(3):424-435. doi: 10.1016/j.pedhc.2024.11.012. Epub 2025 Feb 1. PMID 39891641
- See also: Yorulmaz, D. S., & Kocoglu-Tanyer, D. (2023). A vaccine literacy scale for childhood vaccines: Turkish validity and reliability vaccine literacy scale. Journal of Public Health, 1-9. — https://link.springer.com/article/10.1007/s10389-023-01878-5
- See also: Aharony N, Goldman R, (2017). E-health literacy and the vaccination dilemma: an Israeli perspective. Information Research, 22(2), paper 751. — https://informationr.net/ir/22-2/paper751.html
- See also: Aygün E, Tortop HS, 2020. Ebeveynlerin aşı tereddüt düzeylerinin ve karşıtlık nedenlerinin incelenmesi. Güncel Pediatri, 18(3), 300-16. — https://dergipark.org.tr/en/pub/pediatri/issue/58343/841404
- See also: Rizzi M, Attwell K, Casigliani V, Taylor J, Quattrone F, Lopalco P, 2021. Legitimising a 'zombie idea': childhood vaccines and autism-the complex tale of two judgments on vaccine injury in Italy. International Journal of Law in Context, 1-21. — https://www.cambridge.org/core/journals/international-journal-of-law-in-context/article/legitimising-a-zombie-idea-childhood-vaccines-and-autism-the-complex-tale-of-two-judgments-on-vaccine-injury-in-italy/BF7D7E525FE83898A458202C2D261D66
- See also: Hasar M, Özer ZY, Bozdemir N, 2021. Aşı reddi nedenleri ve aşılar hakkındaki görüşler. Cukurova Medical Journal, 46(1), 166-76. — https://dergipark.org.tr/en/pub/cumj/issue/59504/790733
- See also: Akın B, & Koçoğlu, D. (2017). Randomize kontrollü deneyler. Hacettepe Üniversitesi Hemşirelik Fakültesi Dergisi, 4(1), 73-92. — https://dergipark.org.tr/en/pub/hunhemsire/issue/27606/331915